CLINICAL TRIAL: NCT01319734
Title: Phase 1 Study of Randomized Clinical Trial Comparing Vitamin C Supplementation Plus Oral Hypoglycemic Drugs Versus Hypoglycemic Drugs Alone on Serum Selenium, Zinc, Copper and Malondialdehyde Levels in Type 2 Diabetes Mellitus and Its Microvascular Complications
Brief Title: Vitamin C Supplementation Plus Hypoglycemic Agents Versus Hypoglycemic Agents Alone in Type 2 Diabetes Mellitus
Acronym: Vit C
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Neelain University (Other)
Responsible Party: Principal Investigator, Hamdan Zaki Hamdan, Al-Neelain University, Faculty of Medicine, Department of Biochemistry and Molecular biology, Khartoum, Sudan, Al-Neelain University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Vitamin C; Oxidative stress; Type 2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ascorbic Acid; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C supplementation plus oral hypoglycemic agents arm (Experimental): This group will receive vitamin C supplementation 500mg daily for one month and then assessment will done for the patients.
  Interventions: Dietary Supplement: Vitamin C
- Type 2DM patients receiving oral hypoglycemic agents alone (Active Comparator): this group is the control group who receive oral hypoglycemic agents alone
  Interventions: Drug: glyburide

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C supplementation 500mg
  Arms: Vitamin C supplementation plus oral hypoglycemic agents arm
Drug: glyburide — this group receiving glyburide 5 mg alone
  Arms: Type 2DM patients receiving oral hypoglycemic agents alone

SUMMARY:
Null hypothesis:

No significant effect of vitamin C 500 mg Supplementation on the severity of micro-vascular complications of type 2 Diabetes Mellitus (DM).

Alternative hypothesis:

There is a significant effect of vitamin C 500mg supplementation on the severity of the micro-vascular complications of type 2DM.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 2DM
* patients in good health
* receiving oral hypoglycemic drugs

Exclusion Criteria:

* Insulin dependent diabetes
* receiving vitamin complex
* smoking
* renal disease
* liver disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
improving the renal function | the renal function will be measure at day 1 and after one month
  vitamin c supplementation act as an antioxidants which reduce the oxidative stress and then can improve the renal function.

SECONDARY OUTCOMES:
Vitamin C can improve the visual fields | the visual field will be assesed at day 1 and after one month
  the damage of the eye can be prevented by decreasing the oxidative stress in the eye, this can be accomplished by vitamin C.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdan Z Hamdan, MBBS, MSc, Principal Investigator — Al-Neelain University
Locations (1):
- Jaber abo aliz, Khartoum, Khartoum State, Sudan